CLINICAL TRIAL: NCT03426917
Title: Anesthetic Complication Among Acute Ischemic Stroke Patients During Endovascularization Therapy, Retrospective Descriptive Study
Brief Title: Anesthetic Complication Among Acute Ischemic Stroke Patients During Endovascularization Therapy
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Phuriphong Songarj, Assistant professor, Mahidol University
Other Study IDs: 153/2560(EC1)
Record Dates: First submitted 2018-01-30; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Anesthetic Complication

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective descriptive study

DETAILED DESCRIPTION:
Retrospective chart review from January 2014 to December 2015

ELIGIBILITY:
Inclusion Criteria:

- Acute ischemic stroke patients who received endovascular therapy from January 2015 to December 2016

Exclusion Criteria:

- Age less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - The patients' chart of acute ischemic stroke patients who received endovascular therapy from January 2015 to December 2016
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Anesthetic Complication | Up to 24 hours
  Anesthetic Complication Among Acute Ischemic Stroke Patients During endovascular therapy

CONTACTS AND LOCATIONS:
Overall Officials: Phuriphong Songarj, MD, Principal Investigator — Mahidol University
Locations (1):
- Anesthesiology Department, Bangkok, Thailand